CLINICAL TRIAL: NCT03417518
Title: Effects of General Anesthesia With Propofol Versus Desflurane on Oxidative Stress and Inflammation in Obese Patients Scheduled for Bariatric Surgery
Brief Title: Effects of Anesthesia With Propofol Versus Desflurane in Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B076201420067
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Anesthesia; Obesity
Keywords: Oxidative stress; Bariatric surgery
MeSH Terms: conditions — Obesity | interventions — Desflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desflurane Inhalant Product Group (Active Comparator): general anesthesia with desflurane
  Interventions: Drug: Desflurane Inhalant Product
- Propofol Group (Experimental): general anesthesia with propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane Inhalant Product — General anesthesia will be induced with sufentanyl (0.2µg/kg) and thiopental (5mg/kg) and maintained by desflurane
  Other Names: Suprane
  Arms: Desflurane Inhalant Product Group
Drug: Propofol — General anesthesia will be induced with propofol (2mg/kg) and sufentanyl (0.2µg/kg) and maintained by propofol in a target-controlled infusion mode
  Other Names: Diprivan
  Arms: Propofol Group

SUMMARY:
Evaluate the effects of propofol compared with desflurane on oxidative stress and inflammation markers in obese patients undergoing scheduled bariatric surgery.

DETAILED DESCRIPTION:
Obese patients have a high level of oxidative stress and inflammation activity. Desflurane is an anesthetic gas often used for obese patients. Propofol, another anesthetic agent, has shown an antioxidant property. The aim of the study is to compare the effects of propofol with desflurane on oxidative stress and inflammation markers in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) >35
* scheduled gastric by pass surgery
* American Society of Anesthesiologists (ASA) <III

Exclusion Criteria:

* Allergic to anesthesia agent
* patient refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Malondialdehyde (MDA) level in blood sample | up to 24 hours post bariatric surgery
  Plasma MDA level is measured as an oxidative stress marker before the surgery, at 1 hour, 2 hours, 24 hours post-surgical incision.

SECONDARY OUTCOMES:
C-Reactive Protein (CRP) in blood sample | up to 24 hours post bariatric surgery
  Plasma CRP level is measured as an inflammation marker before the surgery, at 1 hour, 2 hours, 24 hours post-surgical incision.
Monocyte level in blood sample | up to 24 hours post bariatric surgery
  Monocyte level is measured as an inflammation marker before the surgery, at 1 hour, 2 hours, 24 hours post-surgical incision.
Pain assessed by Visual Analog Scale (VAS) | up to 48 hours after surgery
  Pain level is determined at 2 hours, 24 hours and 48 hours post-surgical incision. Visual analog pain score (scale = 0 no pain; 10= worst pain imaginable)
Side-effects (nausea, vomiting, somnolence, respiratory depression) | up to 48 hours after surgery
  Evaluation at 2 hours, 24 hours and 48 hours post-surgical incision

CONTACTS AND LOCATIONS:
Overall Officials: Panayota Kapessidou, Study Director — University Hospital Saint-Pierre (CHU Saint-Pierre), Universite libre de Bruxelles (ULB); Livia Di Marco, doctor, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skalicky J, Muzakova V, Kandar R, Meloun M, Rousar T, Palicka V. Evaluation of oxidative stress and inflammation in obese adults with metabolic syndrome. Clin Chem Lab Med. 2008;46(4):499-505. doi: 10.1515/CCLM.2008.096. PMID 18298345
- [Background] Del Rio D, Stewart AJ, Pellegrini N. A review of recent studies on malondialdehyde as toxic molecule and biological marker of oxidative stress. Nutr Metab Cardiovasc Dis. 2005 Aug;15(4):316-28. doi: 10.1016/j.numecd.2005.05.003. PMID 16054557
- [Background] Murphy PG, Myers DS, Davies MJ, Webster NR, Jones JG. The antioxidant potential of propofol (2,6-diisopropylphenol). Br J Anaesth. 1992 Jun;68(6):613-8. doi: 10.1093/bja/68.6.613. PMID 1319189